CLINICAL TRIAL: NCT03529877
Title: An Interventional, Multicenter, Single Arm, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-EB on Epidermolysis Bullosa (EB)
Brief Title: Allogeneic ABCB5-positive Stem Cells for Treatment of Epidermolysis Bullosa
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Granzer Regulatory Consulting & Services (Other); Ticeba GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: allo-APZ2-EB-II-01
Record Dates: First submitted 2018-04-24; First posted 2018-05-18 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-03

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica; Skin Abnormalities; Congenital Abnormalities; Skin Diseases, Genetic; Somatic Cell Therapy; Mesenchymal Stem Cells; ABCB5; Allogeneic
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa; Skin Abnormalities; Congenital Abnormalities; Skin Diseases, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- allo-APZ2-EB (Experimental): intravenous infusion, three doses of allo-APZ2-EB (2 x 10^6 cells/kg)
  Interventions: Biological: allo-APZ2-EB

INTERVENTIONS:
Biological: allo-APZ2-EB — intravenous infusion of allo-APZ2-EB
  Other Names: allogeneic ABCB5-positive mesenchymal stem cells

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring overall improvement of EB symptoms) and safety (by monitoring adverse events) of three doses of allo-APZ2-EB administered intravenously to patients with recessive dystrophic epidermolysis bullosa (RDEB).

DETAILED DESCRIPTION:
This is an interventional, single arm, non-randomized, open label, phase I/IIa clinical trial to investigate the efficacy and safety of the IMP allo-APZ2-EB in patients with RDEB.

Patients will undergo treatment with the IMP (three repeated intravenous applications) and will be followed up for efficacy for 12 weeks. To assess long-term safety of allo-APZ2-EB one follow-up visit at Month 12 and one follow-up visit at Month 24 post IMP applications is included.

Determination of the EB linked symptoms and quality of life will be assessed by using the EBDASI score, the iscorEB, the change in pain and itch perception, and patient's quality of life in EB. The wound healing process will be documented by photography.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 0 and ≤55 years;

Staggered design for patient enrollment:

1. at least 3 adult patients (safety assessment 2 weeks after last treatment of third patient),
2. at least 3 patients ≥12 to <18 years (safety assessment 2 weeks after first treatment of third patient),
3. at least 3 patients ≥5 to <12 years (safety assessment 2 weeks after first treatment of third patient), and
4. at least 3 patients ≥12 months to <5 years;
5. patients 0 to <12 months (only in the UK);

2. Diagnosed with RDEB (combined diagnosis by genotype assessment [mutation analysis] and correlating phenotype assessment [wound assessment]), patients must have a negative immunofluorescence test result on salt-split skin against proteins of the basement membrane at Visit 1 (existing test results will be accepted);

3. Patient is eligible to participate in this clinical trial based on general health condition at the investigator's discretion;

US only:

Patient is eligible to participate in this clinical trial based on general health condition assessed by specific lab values (Hematology: Absolute neutrophil count >1000/mm3 and platelet count >150,000/mcL; Coagulation: PT and PTT <2x the upper limit of normal for age; Hepatic: AST and ALT <2x the upper limit of normal for age; Renal: Creatinine <2x the upper limit of normal for age; Pulmonary: Oxygen saturation >92% on room air and without supplemental oxygen requirement);

4. Patient/legal representative understands the nature of the procedure and are providing written informed consent prior to any clinical trial procedure;

5. Women of childbearing potential must have a negative urine pregnancy test at Visit 1;

6. Women of childbearing potential and their partner must be willing to use highly effective contraceptive methods during the course of the clinical trial.

Exclusion Criteria:

1. Tumor diseases or history of tumor disease;
2. Known positive result for human immunodeficiency virus 1 and/or 2;
3. Any known allergies to components of the IMP;
4. Evidence of any other medical conditions (such as psychiatric illness or active infection) based on physical examination, or laboratory findings that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment; at investigators discretion;
5. History of prior thrombosis or patients at risk for thrombosis;
6. Clinically significant or unstable concurrent disease or other clinical contraindications (based upon investigator's judgment);
7. Patient/legal representative anticipated to be unwilling or unable to comply with the requirements of the protocol;
8. Pregnant or lactating women;
9. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
10. Previous participation in this clinical trial (except for screening failures due to an exclusion criterion);
11. Known abuse of alcohol, drugs, or medicinal products;
12. Employees of the sponsor, or employees or relatives of the investigator.

Ages: 0 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Overall improvement of EB symptoms after 12 weeks (measured by percentage change of a patient's EBDASI score), score), or last available post-baseline measurement if the Week 12 measurement is missing | Week 12 post baseline, or last available post-baseline measurement if the Week 12 measurement is missing (last observation carried forward [LOCF])
  EBDASI: epidermolysis bullosa disease activity and scarring index; measured in percentage change to baseline score
Assessment of adverse event (AE) occurrence | Up to 24 months
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Overall improvement of EB symptoms after 12 weeks (measured by percentage change of a patient's EBDASI score) | between baseline and week 12 post baseline (without LOCF)
  EBDASI: epidermolysis bullosa disease activity and scarring index; measured in percentage change to baseline score
Overall improvement of EB symptoms after 12 weeks (measured by percentage change of patient's iscorEB), or last available post-baseline measurement if the Week 12 measurement is missing | Week 12 post baseline, or last available post-baseline measurement if the Week 12 measurement is missing (LOCF);
  iscorEB: instrument for scoring clinical outcome of research for epidermolysis bullosa; measured in percentage change to baseline score
Overall improvement of EB symptoms after 12 weeks (measured by percentage change of patient's iscorEB) | between baseline and week 12 post baseline (without LOCF)
  iscorEB: instrument for scoring clinical outcome of research for epidermolysis bullosa; measured in percentage change to baseline score
Overall improvement of EB symptoms at Day 17 (measured by percentage change of a patient's EBDASI score) | between baseline and day 17 post baseline
  EBDASI: epidermolysis bullosa disease activity and scarring index; measured in percentage change to baseline score
Overall improvement of EB symptoms at Day 17 (measured by percentage change of a patient's iscorEB) | between baseline and day 17 post baseline
  iscorEB: instrument for scoring clinical outcome of research for epidermolysis bullosa; measured in percentage change to baseline score
Overall improvement of EB symptoms at Day 35 (measured by percentage change of a patient's EBDASI score) | between baseline and day 35 post baseline
  EBDASI: epidermolysis bullosa disease activity and scarring index; measured in percentage change to baseline score
Overall improvement of EB symptoms at Day 35 (measured by percentage change of a patient's iscorEB) | between baseline and day 35 post baseline
  iscorEB: instrument for scoring clinical outcome of research for epidermolysis bullosa; measured in percentage change to baseline score
Inflammation (measured by panel of inflammation markers) | between baseline and day 17, day 35 and week 12 post baseline
  A panel of inflammation markers will be measured and evaluated.
Pain assessment as per NRS | between baseline and day 17, day 35 and week 12 post baseline
  Pain assessment as per numerical rating scale (NRS) will be evaluated.
Itch assessment as per NRS | between baseline and day 17, day 35 and week 12 post baseline
  Itch assessment as per numerical rating scale (NRS) will be evaluated.
Differences in patient's quality of life in EB | between baseline and day 17, day 35 and week 12 post baseline
  Assessment of quality of life data using an EB-specific quality of life questionnaire
Physical examination until Week 12; | At Screening, baseline, day 17, day 35 and week 12
  A full physical examination will be performed and abnormal physical examination results will be evaluated and reported as AEs.
Vital signs: Body temperature until Week 12; | At Screening, baseline, day 17, day 35 and week 12
  Body temperature will be evaluated at Screening, baseline, day 17, day 35 and week 12
Vital signs: Blood pressure until Week 12; | At Screening, baseline, day 17, day 35 and week 12
  Blood pressure will be evaluated at Screening, baseline, day 17, day 35 and week 12
Vital signs: Heart rate until Week 12; | At Screening, baseline, day 17, day 35 and week 12
  Heart rate will be evaluated at Screening, baseline, day 17, day 35 and week 12
Overall survival at month 24 | month 24 post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Tolar, MD, PhD, Principal Investigator — University of Minnesota, Masonic Cancer Center and Medical Center
Locations (6):
- University of Minnesota, Masonic Cancer Center and Medical Center, Minneapolis, Minnesota, United States
- EB-Haus Austria; Salzburger Landeskliniken (SALK); Paracelsus Medizinische Privatuniversität Salzburg (PMU), Salzburg, Austria
- Hôpital Saint-Louis; Département de dermatologie, Paris, France
- Department of Dermatology, Medical Center-University of Freiburg, Freiburg im Breisgau, Germany
- United Kingdom (2):
  - King's College London; St John's Institute of Dermatology;, London
  - Great Ormond Street Hospital; Dermatology Department, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dieter K, Niebergall-Roth E, Daniele C, Fluhr S, Frank NY, Ganss C, Kiritsi D, McGrath JA, Tolar J, Frank MH, Kluth MA. ABCB5+ mesenchymal stromal cells facilitate complete and durable wound closure in recessive dystrophic epidermolysis bullosa. Cytotherapy. 2023 Jul;25(7):782-788. doi: 10.1016/j.jcyt.2023.01.015. Epub 2023 Mar 1. PMID 36868990
- [Derived] Kiritsi D, Dieter K, Niebergall-Roth E, Fluhr S, Daniele C, Esterlechner J, Sadeghi S, Ballikaya S, Erdinger L, Schauer F, Gewert S, Laimer M, Bauer JW, Hovnanian A, Zambruno G, El Hachem M, Bourrat E, Papanikolaou M, Petrof G, Kitzmuller S, Ebens CL, Frank MH, Frank NY, Ganss C, Martinez AE, McGrath JA, Tolar J, Kluth MA. Clinical trial of ABCB5+ mesenchymal stem cells for recessive dystrophic epidermolysis bullosa. JCI Insight. 2021 Nov 22;6(22):e151922. doi: 10.1172/jci.insight.151922. PMID 34665781
- [Derived] Kerstan A, Niebergall-Roth E, Esterlechner J, Schroder HM, Gasser M, Waaga-Gasser AM, Goebeler M, Rak K, Schrufer P, Endres S, Hagenbusch P, Kraft K, Dieter K, Ballikaya S, Stemler N, Sadeghi S, Tappenbeck N, Murphy GF, Orgill DP, Frank NY, Ganss C, Scharffetter-Kochanek K, Frank MH, Kluth MA. Ex vivo-expanded highly pure ABCB5+ mesenchymal stromal cells as Good Manufacturing Practice-compliant autologous advanced therapy medicinal product for clinical use: process validation and first in-human data. Cytotherapy. 2021 Feb;23(2):165-175. doi: 10.1016/j.jcyt.2020.08.012. Epub 2020 Oct 1. PMID 33011075